CLINICAL TRIAL: NCT05256004
Title: Association of Cardiac Biomarkers of Heart Failure and Iron Status in Hemodialysis Patients
Brief Title: Cardiac Biomarkers and Iron Status in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 110070
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure; Iron-deficiency
Keywords: Heart failure; Iron status; Cardiac biomarkers
MeSH Terms: conditions — Heart Failure; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Peripheral arterial disease (PAD) a condition characterized by atherosclerotic occlusive disease of the lower extremities is commonly observed in patients with chronic kidney disease (CKD) patients, particularly those on dialysis. We conducted detailed biomarkers such as thrombospondin and related inflammatory biomarkers for the risk of developing and presence of PAD. Thrombospondin-4 (TSP-4) is an extracellular matrix protein of the vessel wall. Despite bench evidence, its significance in the clinical setting of chronic kidney disease (CKD) is missing

Methods:

This is a cross-sectional, single-center study. A cohort of 450 patients aged 20 or over, who have been on HD for at least 3 months prior to enrollment (Dec 1, 2021) will be included. TSP-4 and TSP-1 will be measured in HD patients using a commercially available ELISA. PAD is diagnosed by the ankle-brachial index (ABI) We will measure related blood biomarkers such as serum hs-cTnT, N-terminal probrain natriuretic peptide, s-Klotho and FABP-4.

DETAILED DESCRIPTION:
Study Population and Data Source

This is a cross-sectional, single-center study which will be conducted in the Dialysis Center of Tungs' Taichung MetroHarbor Hospital (TTMHH) in the coastal region of central Taiwan. A cohort of 500 patients aged 20 or over, who have been on HD for at least 3 months prior to enrollment will be included. The medical charts of these patients are reviewed for eligibility identification, and should be compatible with the inclusion/exclusion criteria and enrolled in our analysis. The research was conducted ethically in accordance to the World Medical Association Declaration of Helsinki. Subjects provided written informed consent and the Local Ethical Committee approved the study.

The baseline data such as demographics, comorbidities, anthropometrics, and relevant laboratory data, clinical diagnosis of hear failure based on cardiac echocardiograhy measurements, and medication history will be collected. None of the patients were receiving blood transfusions, or intravenous iron therapy within two weeks before the time of inclusion. Doppler echocardiography using standardized equipment and complying with recommendations from the American Society of Echocardiography (2009)[20]. The biplane method of disks was used to measure left ventricular (LV) EF. Patients were eligible for the study if they had the New York Heart Association (NYHA) functional class II-IV; HFrEF and left ventricular EF (LVEF)≤40%. The characteristics of patients will be exclude from our study were (1) decompensated cirrhosis , (2) neoplastic diseases , (3) incomplete data, (4) receiving hemodialysis < 3 months and active infection.

Iron Status and Other Laboratory Measurements

Blood was drawn with EDTA anticoagulant in the morning after an overnight fast of at least 12 h before a dialysis session. The samples were separated via centrifugation (3000 rpm, 10 min) and immediately stored at -80°C for subsequent assays. Glucose, high-density lipoprotein cholesterol HDL), triglycerides and total cholesterol are all measured by standard assays using the analyzer. Low-density lipoprotein cholesterol (LDL) is measured by standard assay. High-sensitivity C-reactive protein (hsCRP) and are measured using standard nephelometry. Serum hs-cTnT was measured using a sandwich immunoassay method, a novel highly sensitive assay with a lower measurable limit of 3 ng/L.

Iron deficiency was defined using the Kidney Disease Outcomes Quality Initiative guidelines criteria: ferritin < 100 ng/mL or transferrin saturation (TSAT) < 20% when ferritin is < 800 ng/mL.[21] Serum iron was measured using spectrophotometry; serum ferritin and transferrin were measured using immunoturbidimetry. The TSAT was estimated using the formula: TSAT serum iron (μg/dL)/[serum transferrin (mg/dL)×1.25].[22] Additional measures of iron status were: serum soluble transferrin receptor (sTfR) (measured using an enzyme immunoassay),[23-24] and ferritin index. Ferritin index has been proposed as a useful tool in the diagnosis of ID states, where ratios > 2 suggest ID. The ferritin index is calculated by dividing sTfR (expressed in nmol/L or mg/L) by log10 ferritin (measured in ng/mL) and is thus increased whenever sTfR is raised and or ferritin is reduced.[25] Hepcidin is a 25-amino-acid peptide that is produced mainly by the liver, secreted into plasma, and excreted in urine. It is the main regulator of systemic iron homeostasis which restricts the intestinal iron absorption and iron release from macrophages [26]. Serum hepcidin was assayed using a hepcidin ELISA Kit(Human Hepc25), a sandwich-ELISA technique.

Measurement of biomarkers

The GDF15 concentrations are determined by a quantitative sandwich enzyme immunoassay technique (Quantikine®; R&D Systems, Inc. Minneapolis, MN, USA). Quality control (QC) samples from R&D Systems, which had a total coefficient of variation (CV) of 6.3% at low concentrations (159 ng/L), 9.7% at medium concentrations (436 ng/L), and 15.1% at high concentrations (827 ng/L), were included in each assay and results were accepted when QCs fell within manufacturer-specified lot-specific concentration. Overall range of GDF15 detection was 308-13790 ng/L. Gal-3 concentration in plasma was analyzed in duplicate by a commercially available ELISA kit (Norcross, GA or BG Medicine, Inc., Waltham, Mass., USA). Soluble ST2 levels were assessed on baseline samples using a highly sensitive sandwich monoclonal immunoassay (Presage® ST2 Assay, Critical Diagnostics, New York, NY), with a lower limit of detection of 2 ng/mL, an upper limit of detection of 200 ng/mL, an intra-assay coefficient of variation <2.5%, and an interassay coefficient of variation of<4.6%15. Serum H-FABP was measured by an enzyme-linked immunosorbent assay (Hycult Biotech, Uden, the Netherlands). The hsTnT concentrations was measured by electro-chemiluminescence immunoassay using the troponin T high-sensitivity assays, on a Cobas analyser (Roche Diagnostics GmbH, Mannheim, Germany or Abott ). Serum NT-pro-BNP was analyzed using a commercial NT-proBNP ELISA kit. Detection of NT-proBNP ranged from 12 ng/L to 35 000 ng/L and hsTnT ranged between 3 ng/L and 1172 ng/L. All assays were performed in duplicate by technicians blinded to the all clinical data.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes aged 20 years or over
2. Received stable hemodialysis at least 3 months.
3. Written informed consent.

Exclusion Criteria:

1. decompensated cirrhosis.
2. neoplastic diseases.
3. incomplete data.
4. receiving hemodialysis < 3 months and active infection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients have to be at least 20-years-old and on outpatient hemodialysis (HD) for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Measures of iron status | 1 years
  indicating iron storage (ferritin), iron transport (transferrin saturation), regulator of systemic iron homeostasis (hepcidin) and iron demand (soluble transferrin receptor) ,Iron dysmetabolism potentially contributes to heart failure

SECONDARY OUTCOMES:
Analysis of biomarkers of GDF-15 | 1 years
  The GDF-15 was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of Galectin-3 | 1 years
  The Galectin-3 was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of Soluble ST2 | 1 years
  The Soluble ST2 was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of hs-cTnT | 1 years
  The hs-cTnT was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of N-terminal probrain natriuretic peptide | 1 years
  The N-terminal probrain natriuretic peptide was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Analysis of biomarkers of FABP-4 | 1 years
  The FABP-4 was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan